CLINICAL TRIAL: NCT04028986
Title: Efficacy of Ulipristalacetate in Comparison to Surgery Before IVF/ICSI-treatment in Women With Intramural Fibroids: Effect on Reproductive Outcome.
Brief Title: Esmya Versus Surgery Before IVF/ICSI
Status: Active, not recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Stefan Cosyns, Principal Investigator, Universitair Ziekenhuis Brussel
Other Study IDs: B.U.N.14320152
Record Dates: First submitted 2019-07-15; First posted 2019-07-23 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Fibroid; Uterus Tumor, Complicating Pregnancy; Infertility, Female; Surgical Procedure, Unspecified
Keywords: ulipristalacetate; fertility treatment; IVF/ICSI; fibroid
MeSH Terms: conditions — Leiomyoma; Uterine Neoplasms; Pregnancy Complications; Infertility, Female | interventions — ulipristal acetate; Tablets; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery group: patients treated by surgery before starting the IVF/ICSI treatment
- Ulipristalacetate group: patients treated by ulipristalacetate before starting IVF/ICSI treatment
  Interventions: Drug: Ulipristal Acetate 5 MG Oral Tablet

INTERVENTIONS:
Drug: Ulipristal Acetate 5 MG Oral Tablet — use of ulipristalacetate OR surgery before fertility treatment
  Other Names: surgery for fibroid
  Groups: Ulipristalacetate group

SUMMARY:
Studying the possible outcome differences between surgery or medical treatment with ulipristalacetate (UPA) solely before 'in-vitro fertilisation/intracytoplasmic sperm injection' (IVF/ICSI) treatment in infertile couples.

DETAILED DESCRIPTION:
Uterine fibroids are the most common benign uterine tumors in women of reproductive age. Symptoms are depending on size, number and localisation of the fibroids. Heavy menstrual bleeding, anaemia, abdominal pain, dyspareunia and urinary symptoms are often put forward.

Intramural and especially submucous myomas are known to decrease fertility and augment miscarriage rate. Some studies have demonstrated a negative effect of intramural fibroids on fertility outcome, while others do not. A recent meta-analysis found adverse pregnancy outcomes associated not only with submucous and intramural fibroids distorting the uterine cavity, but also with intramural fibroids not distorting the cavity.

Ulipristalacetate (Esmya®) is currently used to pre-treat symptomatic women with fibroids before surgical intervention. Esmya® has been demonstrated to be safe and effective in the treatment of fibroids. Due to apoptosis sometimes a reduction in volume of the myoma is seen. This effect could influence the fertility and operative outcome.

Current options are available before assisted reproductive technology (ART) for infertile women diagnosed with fibroids:

1. no treatment
2. medical pre-treatment before ART:

   1. with gonadotropin-releasing hormone (GnRH)-analogues followed by controlled ovarian stimulation
   2. with ESMYA followed by controlled ovarian stimulation
3. surgical treatment after medical pre-treatment before ART:

   1. after pre-treatment with GnRH analogues followed by myomectomy
   2. after ESMYA followed by myomectomy
4. surgical treatment without medical pre-treatment

In our tertiary infertility centre, at the discretion of the physician, as well ESMYA treatment solely or surgery before starting an IVF/ICSI treatment in women with intramural fibroids are often used. Is there a difference in ongoing pregnancy rate after IVF/ICSI in these patients?

Objective of the study Prospective and retrospective gathering of information regarding the efficacy of IVF/ICSI treatment (ongoing pregnancy rates) in patients undergoing medical or surgical treatment preceding their IVF/ICSI treatment in case of diagnosis of intramural fibroids. Especially ongoing pregnancy rates between patients receiving the ESMYA solely treatment and patients pre-treated by myomectomy before IVF/ICSI will be studied once sufficient data have been collected to deduce valuable study results.

ELIGIBILITY:
Inclusion Criteria:

* 1st, 2nd or 3th IVF/ICSI attempt
* infertility Indications:

  * unexplained
  * tubal
  * male/donor sperm
  * endometriosis I/II
* Body Mass Index (BMI) >18 - < 30
* Basal Follicle Stimulating Hormone (FSH) < 10 IU/L
* anti-mullerian hormone (AMH) > 1 ng/ml
* Normal ultrasound apart from the following:

  * Type 2 fibroid : ≤2cm diameter
  * Type 3 - 5 fibroids: with diameter ≥ 3 and ≤10cm according to classification of European Society for Gynecological Endoscopy (ESGE )

Exclusion Criteria:

* More than 2 submucous fibroids
* Poor responders
* Severe male factor

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: females with fibroids and infertility
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
ongoing pregnancy rates | 2 years

SECONDARY OUTCOMES:
Miscarriage rate | 2 years
Time to pregnancy | 2 years
  years
Obstetric outcome described as live birth | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis UZBrussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No